CLINICAL TRIAL: NCT02442167
Title: Fluorescence in Situ Hybridization (FISH) Improves Performance of Conventional Cytology for the Diagnosis of Malignant Biliary Tract Strictures in Thai Patients
Brief Title: Performance of FISH for the Diagnosis of Malignant Biliary Strictures in Thai Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Lewis R. Roberts, PI, Mayo Clinic
Other Study IDs: 14-008579
Record Dates: First submitted 2015-05-06; First posted 2015-05-13 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Bile Duct Stricture; Malignancy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Brush samples obtained from endoscopic retrograde cholangiopancreatography
Oversight: Data Monitoring Committee: No

SUMMARY:
Fluorescence in situ hybridization (FISH) has improved the diagnostic performance of cytology for evaluation of malignant biliary strictures in the US and Europe. The utility of FISH for diagnosis of biliary strictures in Asia is currently unknown. The investigators conducted a prospective study in 2 university hospitals to determine diagnostic performance of FISH for the diagnosis of malignant biliary strictures in Thai patients.

DETAILED DESCRIPTION:
Fluorescence in situ hybridization (FISH) has improved the diagnostic performance of cytology for evaluation of malignant biliary strictures in the US and Europe. The utility of FISH for diagnosis of biliary strictures in Asia is currently unknown. The investigators aimed to compare the sensitivity of FISH and conventional cytology for the diagnosis of malignant biliary strictures in Thai patients. A prospective study was performed in 2 university hospitals between 2010 and 2013. Patients being evaluated for malignant-appearing biliary strictures were included. Bile duct brushings were collected and assessed by cytology and FISH. Sensitivities with 95% confidence intervals of cytology and FISH were main outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical suspicion of malignant biliary tract strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated for malignant appearing biliary tract strictures who undergo ERCP
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sensitivities with 95% confidence intervals of FISH | Up to 12 months
  Sensitivities with 95% confidence intervals of FISH and routine cytology will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Lewis R Roberts, MB, ChB, PhD, Principal Investigator — Mayo Clinic, Rochester, MN, USA